CLINICAL TRIAL: NCT06640920
Title: A Phase 1 Randomized, Double-Blind Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Bioavailability of NSI-8226 in Healthy Participants
Brief Title: A Study to Investigate Efficacy and Safety of NSI-8226 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Uniquity One (UNI) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSI-8226-101
Record Dates: First submitted 2024-09-13; First posted 2024-10-15 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A (Experimental): NSI-8226
  Interventions: Biological: Cohort A
- Cohort B (Experimental): NSI-8226
  Interventions: Biological: Cohort B
- Cohort C (Experimental): NSI-8226
  Interventions: Biological: Cohort C
- Cohort D (Experimental): NSI-8226
  Interventions: Biological: Cohort D

INTERVENTIONS:
Biological: Cohort A — Administered IV High dose
  Arms: Cohort A
Biological: Cohort B — Administered SC Low Dose
  Arms: Cohort B
Biological: Cohort C — Administered SC Mid Dose
  Arms: Cohort C
Biological: Cohort D — Administered SC High Dose
  Arms: Cohort D

SUMMARY:
A Phase 1 Randomized, Double-Blind Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Bioavailability of NSI-8226 in Healthy Participants.

ELIGIBILITY:
Key Inclusion Criteria:

1. At the time of initial screening, in general good health (age 18 to 65 years);

Key Exclusion Criteria:

1. Pregnancy or breastfeeding during the study.
2. Chronic infection - Treatment with prohibited medications.
3. Treatment with prohibited medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 140 days
  To evaluate the incidence of treatment emergent adverse events of NSI-8826 in healthy participants according to Common Terminology Criteria for Adverse Events (CTCAE) V4.0

SECONDARY OUTCOMES:
Absolute bioavailability | 140 days
  Pharmacokinetics (PK) and absolute bioavailability of NSI-8226 in healthy participants.
Concentration of immunogenicity | 140 days
  Immunogenicity profile of NSI-8226 in healthy participants.
Parameters in healthy participants | 140 days
  Pharmacodynamic (PD) parameters of NSI-8226 in healthy participants.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Lee, MD, Study Chair — Vice President, Clinical Research
Locations (1):
- Research Site, Cincinnati, Ohio, United States